CLINICAL TRIAL: NCT06915194
Title: SMART Pilot Trial of Glycemic Screening Outreach
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kenrik Duru, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: IRB-24-6330
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-04

CONDITIONS: Overweight (BMI > 25); Obesity
Keywords: diabetes screening
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Initial text, follow-up text, letter (Experimental): Participants are initially randomized to glycemic screening invitations by text, and then if they are not screened within 30 days, then they are re-rerandomized to another glycemic screening invitation by text. If they are still not screened in another 30 days then they receive a mailed letter encouraging glycemic screening.
  Interventions: Behavioral: Text message; Behavioral: Mailed letter
- Initial portal, follow-up portal, letter (Experimental): Participants are initially randomized to glycemic screening invitations by patient portal, and then if they are not screened within 30 days, then they are re-rerandomized to another glycemic screening invitation by patient portal. If they are still not screened in another 30 days then they receive a mailed letter encouraging glycemic screening.
  Interventions: Behavioral: Patient portal message; Behavioral: Mailed letter
- Initial text, follow-up portal, letter (Experimental): Participants are initially randomized to glycemic screening invitations by text, and then if they are not screened within 30 days, then they are re-rerandomized to another glycemic screening invitation by patient portal. If they are still not screened in another 30 days then they receive a mailed letter encouraging glycemic screening.
  Interventions: Behavioral: Text message; Behavioral: Patient portal message; Behavioral: Mailed letter
- Initial portal, follow-up text, letter (Experimental): Participants are initially randomized to glycemic screening invitations by patient portal, and then if they are not screened within 30 days, then they are re-rerandomized to another glycemic screening invitation by text. If they are still not screened in another 30 days then they receive a mailed letter encouraging glycemic screening.
  Interventions: Behavioral: Text message; Behavioral: Patient portal message; Behavioral: Mailed letter
- Usual care (No Intervention): Patients do not receive any glycemic screening invitations

INTERVENTIONS:
Behavioral: Text message — Participants receive a text message encouraging glycemic screening
  Arms: Initial portal, follow-up text, letter; Initial text, follow-up portal, letter; Initial text, follow-up text, letter
Behavioral: Patient portal message — Participants receive a patient portal message encouraging glycemic screening
  Arms: Initial portal, follow-up portal, letter; Initial portal, follow-up text, letter; Initial text, follow-up portal, letter
Behavioral: Mailed letter — Participants receive a mailed letter encouraging glycemic screening
  Arms: Initial portal, follow-up portal, letter; Initial portal, follow-up text, letter; Initial text, follow-up portal, letter; Initial text, follow-up text, letter

SUMMARY:
Approximately 130 million Americans have prediabetes or type 2 diabetes (T2D) but remain unscreened and/or unaware of their diagnosis. While prediabetes/T2D screening, also known as glycemic screening, is endorsed in national guidelines, there is almost no research on how to increase screening rates, or evaluations of interventions testing the effectiveness of screening promotion strategies. The American Medical Association has published prediabetes quality measures that apply to UCLA Health as well as all other health systems, specifically tracking the percentage of adult patients with risk factors for T2D due for glycemic screening for whom the screening process was initiated. However, there is no current systemic effort underway at UCLA, or most other health systems, to encourage glycemic screening. We are proposing a pilot trial of the first SMART (Sequential Multiple Assignment Randomized Trial) for glycemic screening. Our SMART experiment will provide preliminary feasibility and acceptability data for a larger, multisite trial that will provide vital guidance to optimize screening approaches for a growing number of screening-eligible patients so that they may seek earlier detection, treatment, and/or access to lifestyle programs and interventions for T2D or prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese

Exclusion Criteria:

* Existing type 2 diabetes, A1c drawn within past 3 years

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 90 days
  Receipt of hemoglobin A1c screening for dysglycemia

SECONDARY OUTCOMES:
Acceptability survey | 90 days
  Participants will receive a Qualtrics survey with the following 5 items:
  1. How did you feel about the messages recommending that you come in for a blood test to check your hemoglobin A1c (blood sugar) level?
  2. How clear were the messages recommending that you come in for a blood test to check your hemoglobin A1c (blood sugar) level?
  3. Did the messages affect the chances that you would get the hemoglobin A1c (blood sugar) level?
  4. Did the messages cause you any anxiety or stress?
  5. How concerned were you that the messages were from scammers not associated with UCLA?

CONTACTS AND LOCATIONS:
Overall Officials: Obidiugwu K Duru, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We may or may not attempt to publish this pilot trial